CLINICAL TRIAL: NCT03514186
Title: The Intensive Comprehensive Aphasia Program (ICAP): A Randomized Clinical Trial
Brief Title: The Intensive Comprehensive Aphasia Program (ICAP)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shirley Ryan AbilityLab (Other)
Collaborators: Northwestern University (Other)
Responsible Party: Principal Investigator, Leora Cherney, Scientific Chair, Think & Speak Lab, Shirley Ryan AbilityLab
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 81035
Record Dates: First submitted 2018-04-17; First posted 2018-05-02 (Actual); Last update posted 2022-06-21 (Actual); Status verified 2022-06

CONDITIONS: Aphasia; Stroke
Keywords: Aphasia; Speech and Language Treatment; ICAP; Intensive Comprehensive Aphasia Program
MeSH Terms: conditions — Aphasia; Stroke; Speech | interventions — Speech Therapy

STUDY DESIGN:
Intervention Model Description: Both treatment arms will provide 60 hours of comprehensive aphasia therapy. In the ICAP arm, the 60 hours of treatment will be applied intensively, 4 hours per day, 5 days a week for three weeks. In the Distributed Treatment arm, the 60 hours of comprehensive treatment will be distributed over 15 weeks (i.e. two 2-hour visits per week).
Who Masked: Outcomes Assessor
Masking Description: Because of the nature of the intervention, neither the treating SLPs nor the subjects can be masked regarding the scheduling of treatment. To minimize outcome ascertainment bias, an evaluator (testing speech-language pathologist) who is not directly associated with the daily activities of the trial and, therefore, blind to the treatment arm will administer and score all the assessments. Subjects will be introduced to the treatment arm to which they have been assigned with a script that emphasizes similar expectations from the intervention, regardless of the treatment group. This will reduce subject bias resulting from such beliefs that one of the therapies is less effective.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intensive Comprehensive Aphasia Program (Experimental): 60 hours of comprehensive speech and language therapy applied intensively, 4 hours per day, 5 days a week for three weeks.
  Interventions: Behavioral: Speech and Language Therapy
- Distributed Comprehensive Aphasia Tx (Active Comparator): 60 hours of comprehensive speech and language therapy distributed over 15 weeks (i.e. two 2-hour visits per week).
  Interventions: Behavioral: Speech and Language Therapy

INTERVENTIONS:
Behavioral: Speech and Language Therapy — Includes:
  * one hour of individual therapy using a multimodality treatment called Verb Network Strengthening Treatment (VNeST) that simultaneously targets semantics (word retrieval) and syntax (sentence construction);
  * one hour of constraint induced language therapy (CILT) where participants are paired and practice requesting and providing specific information using only spoken language;
  * one hour in the computer lab working on programs called Oral Reading for Language in Aphasia (ORLA) and AphasiaScripts; and
  * one hour in a conversation group that emphasizes multimodality communication

SUMMARY:
The purpose of this study is to conduct a randomized clinical trial that assesses the efficacy and cost-effectiveness of an Intensive Comprehensive Aphasia Program (ICAP), specifically focusing on the variable of intensity. Half of the participants will receive 60 hours of intensive treatment over three weeks, while the other half will receive the same amount and type of comprehensive treatment distributed over 15 weeks.

DETAILED DESCRIPTION:
Recent research has emphasized the need for intensive aphasia treatment in order to make the long-term neuroplastic changes associated with recovery and rehabilitation following a stroke. Furthermore, studies have indicated that intensive aphasia treatment is more efficacious than less intensive treatment. Rather than being influenced by such evidence, the reality is that public and private payers are drastically reducing services to persons with aphasia (PWA). Legislation has seriously curtailed the amount of treatment a PWA may receive after hospitalization. Often patients are eligible for only a limited number of treatment sessions over a limited period of time. In some cases, they may not receive any treatment for their communication disorder following their acute hospitalization. Reduced resources (e.g. transportation difficulties, therapist shortages in rural areas) also may severely limit available services.

The Intensive Comprehensive Aphasia Program (ICAP) may be a creative, cost-effective and sustainable option for delivering meaningful and necessary aphasia services. Despite the growing numbers of ICAPs, there is little evidence about their efficacy, effectiveness, or cost-effectiveness. All stakeholders need this evidence. Funding agencies require evidence to make decisions about their investments in aphasia rehabilitation. People with aphasia and their families should have evidence prior to investing their money and time into such programs, and speech and language pathologists have an ethical obligation to provide evidence-based practices.

Based on evidence regarding treatment intensity that has translated principles of neuroplasticity from animal models to stroke recovery, the investigators hypothesize that 60 hours of comprehensive treatment will result in significant improvements in (a) performance-based, (b) client-reported, and (c) surrogate-reported assessments of communication skills, community participation, and health-related quality of life. They also hypothesize that when 60 hours of comprehensive treatment is provided intensively over 3 weeks, the magnitude and rate of improvement as well as the extent to which improvements are maintained will be greater than when the 60 hours of comprehensive treatment is distributed over 15 weeks. Because the investigators hypothesize that the magnitude and rate of improvement will be greater with the intensive ICAP than with the distributed ICAP, they further hypothesize that the intensive ICAP will be more cost-effective than the distributed ICAP.

ELIGIBILITY:
Inclusion Criteria:

1. diagnosis of an aphasia subsequent to a left-hemisphere infarct that is confirmed by CT scan or MRI
2. an Aphasia Quotient score on the Western Aphasia Battery of 20-85.
3. 6 months post injury
4. premorbidly fluent in English
5. receiving no concomitant speech-language therapy

Exclusion Criteria:

1. diagnosis of Global aphasia
2. any other neurological condition (other than cerebral vascular disease) that could potentially affect cognition or speech, such as Parkinson's Disease, Alzheimer's disease and other dementias, or traumatic brain injury
3. any significant psychiatric history prior to the stroke, such as severe major depression or psychotic disorder requiring hospitalization (subjects with mood disorders who are currently stable on treatment will be considered)
4. active substance abuse.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2015-07-15 (Actual); Primary Completion 2019-03 (Actual); Study Completion 2022-06 (Actual)

PRIMARY OUTCOMES:
Language Quotient of the Western Aphasia Battery-Revised (WAB-R LQ) | Change from pre-treatment to post-treatment (i.e. following completion of 60 hours of treatment at 3 weeks or 15 weeks depending on group assignment)
  Includes a measure of auditory comprehension, oral expression, reading and written expression skills. Change from baseline to post-treatment and follow-up is reported.

SECONDARY OUTCOMES:
Language Quotient of the Western Aphasia Battery-Revised (WAB-R LQ) | Change from pre-treatment to 3 month follow-up
  Includes a measure of auditory comprehension, oral expression, reading and writing
Assessment for Living with Aphasia (ALA) | Change from pre-treatment to post-treatment (i.e. following completion of 60 hours of treatment at 3 weeks or 15 weeks depending on group assignment)
  A pictographic self-report measure designed to assess outcomes associated with the impact of aphasia on daily life.
Assessment for Living with Aphasia (ALA) | Change from pre-treatment to 3 month follow-up
  A pictographic self-report measure designed to assess outcomes associated with the impact of aphasia on daily life.
The Communication Confidence Rating Scale for Aphasia (CCRSA) | Change from pre-treatment to post-treatment (i.e. following completion of 60 hours of treatment at 3 weeks or 15 weeks depending on group assignment)
  Self-reported measure that assesses perceived confidence in a variety of different communication situations and with different people. Scores range from 0 - 40, with higher scores indicating greater perceived confidence.
The Communication Confidence Rating Scale for Aphasia (CCRSA) | Change from pre-treatment to 3 month follow-up
  Self-reported measure that assesses perceived confidence in a variety of different communication situations and with different people. Scores range from 0 - 40, with higher scores indicating greater perceived confidence.
The Communicative Effectiveness Index (CETI) | Change from pre-treatment to post-treatment (i.e. following completion of 60 hours of treatment at 3 weeks or 15 weeks depending on group assignment)
  A proxy-reported 16 visual analogue scale items that assess areas of functional communication in the participant's living environment. Scores range from 0 - 100, with higher scores indicating better communication effectiveness.
The Communicative Effectiveness Index (CETI) | Change from pre-treatment to 3 month follow-up
  A proxy-reported 16 visual analogue scale items that assess areas of functional communication in the participant's living environment. Scores range from 0 - 100, with higher scores indicating better communication effectiveness.

CONTACTS AND LOCATIONS:
Overall Officials: Leora Cherney, PhD, Principal Investigator — Shirley Ryan AbilityLab
Locations (1):
- Shirley Ryan AbilityLab, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No